CLINICAL TRIAL: NCT00406705
Title: A Randomized Controlled Trial to Study the Effect of Exercise Training Breathing Helium-Hyperoxia on The Exercise Tolerance and Quality of Life of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Breathing Helium-Hyperoxia During Pulmonary Rehabilitation in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSI 824
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Lung Diseases; Bronchitis, Chronic
Keywords: Exercise Tolerance; Dyspnea; Rehabilitation; Helium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Lung Diseases; Bronchitis, Chronic; Dyspnea

INTERVENTIONS:
Behavioral: Helium-Hyperoxia

SUMMARY:
The purpose of this study is to examine whether breathing helium-hyperoxia during exercise in a pulmonary rehabilitation program can improve the exercise tolerance and health related quality of life of patients with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
It is well accepted that the exercise training as part of a comprehensive pulmonary rehabilitation program can improve exercise tolerance, functional status and quality of life in patients with COPD. It is feasible that if patients were able to perform a greater volume or intensity of exercise during rehabilitation then the outcomes of the program would be improved. Recent research has demonstrated that breathing a helium-hyperoxic gas mixture can significantly reduce dynamic hyperinflation and dyspnea during exercise in patients with COPD and can increase exercise tolerance to a greater extent than breathing room air or a nitrogen-based hyperoxic gas. If patients with COPD were to breathe a helium-hyperoxic gas during exercise they should be able to tolerate a greater intensity of exercise while maintaining similar levels of exertional symptoms to those observed at lower exercise intensities breathing room air. As a result patients randomized to the helium-hyperoxia condition should obtain greater improvements in exercise tolerance than those receiving usual care (i.e. breathing room air)

Comparisons: Standard pulmonary rehabilitation of patients with COPD receiving either usual care (air breathing) or helium-hyperoxia (40% O2, 60% Helium).

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC<70% predicted;
* FEV1<70% predicted;
* RV>140% predicted.

Exclusion Criteria:

* Cardiovascular contraindications to exercise;
* Musculoskeletal abnormalities that limit exercise tolerance;
* SpO2<85% during a constant work rate test;
* On supplemental oxygen.
* Exacerbation within the last month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Start 2005-03; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Constant-load exercise tolerance after 6 weeks of exercise rehabilitation

SECONDARY OUTCOMES:
Maximum oxygen consumption after 6 weeks of exercise rehabilitation
Quality of Life measured after 6 weeks of exercise rehabilitation
Dyspnea at an isotime during constant-load exercise after 6 weeks of exercise rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Neil D Eves, PhD, Principal Investigator — University of Calgary, AB, Canada
Locations (1):
- Caritas Centre for Lung Health, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Eves ND, Petersen SR, Haykowsky MJ, Wong EY, Jones RL. Helium-hyperoxia, exercise, and respiratory mechanics in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2006 Oct 1;174(7):763-71. doi: 10.1164/rccm.200509-1533OC. Epub 2006 Jul 13. PMID 16840742
- [Derived] Eves ND, Sandmeyer LC, Wong EY, Jones LW, MacDonald GF, Ford GT, Petersen SR, Bibeau MD, Jones RL. Helium-hyperoxia: a novel intervention to improve the benefits of pulmonary rehabilitation for patients with COPD. Chest. 2009 Mar;135(3):609-618. doi: 10.1378/chest.08-1517. Epub 2008 Nov 18. PMID 19017883